CLINICAL TRIAL: NCT07163910
Title: Clinical Study of Homoharringtonine Combined With Androgen Deprivation Therapy in Neoadjuvant Treatment of Prostate Cancer
Brief Title: Homoharringtonine Plus Androgen Deprivation Therapy in the Neoadjuvant Treatment of Prostate Cancer: A Single-Arm Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: baotai Liang (Other)
Collaborators: The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); Subei People's Hospital of Jiangsu Province (Other); The First People Hospital of Nantong City (Unknown)
Responsible Party: Sponsor-Investigator, baotai Liang, lead researcher, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZDSYLL510-P02
Record Dates: First submitted 2025-08-20; First posted 2025-09-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Homoharringtonine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Localized High-Risk/Very High-Risk and Regional Lymph Node-Metastatic Prostate Cancer (Experimental): This study is a single-arm clinical trial, and eligible patients will be enrolled. For the enrolled patients, the treatment regimen will consist of intravenous infusion of 1mg homoharringtonine combined with 250ml of 5% glucose injection, administered once daily for two consecutive days. Patients with localized high-risk/very high-risk prostate cancer or prostate cancer with local lymph node metastasis will receive at least one cycle of the above treatment plus continuous androgen deprivation therapy.All patients will undergo radical prostatectomy within 3 weeks (±7 days) after the completion of treatment.
  Interventions: Drug: homoharringtonine; Procedure: Radical prostatectomy
- Patients with metastatic prostate cancer (Experimental): This study is a single-arm clinical trial, and eligible patients will be enrolled. For the enrolled patients, the treatment will consist of intravenous infusion of 1mg homoharringtonine plus 250ml of 5% glucose injection, administered once daily for two consecutive days. For patients with metastatic prostate cancer, the medication will be repeated after an interval of three weeks following one treatment cycle, with the entire course lasting for at least three cycles, in addition to continuous androgen deprivation therapy. All patients will undergo radical prostatectomy within 3 weeks (±7 days) after the completion of treatment.
  Interventions: Drug: homoharringtonine; Procedure: Radical prostatectomy

INTERVENTIONS:
Drug: homoharringtonine — Intravenous infusion of 1mg homoharringtonine plus 250ml of 5% glucose injection, administered once daily for two consecutive days.
  Other Names: drug therapy
Procedure: Radical prostatectomy — All patients will undergo radical prostatectomy within 3 weeks (±7 days) after the completion of treatment.
  Other Names: operative treatment

SUMMARY:
The project aims to verify the therapeutic effect of neoadjuvant homoharringtonine combined with androgen deprivation therapy in patients with localized high-risk/very high-risk, regional lymph node-metastatic, or metastatic prostate cancer before radical prostatectomy through clinical trials, thereby identifying an effective treatment for patients with advanced prostate cancer.

DETAILED DESCRIPTION:
This study is a single-arm clinical trial, and eligible patients will be enrolled. For the enrolled patients, they will receive an intravenous infusion of homoharringtonine (1 mg) plus an intravenous infusion of 5% glucose injection (250 ml), once daily for two consecutive days. Patients with localized high-risk/very high-risk and regional lymph node-metastatic prostate cancer will receive at least one cycle of the above treatment plus continuous androgen deprivation therapy; patients with metastatic prostate cancer will receive one cycle of treatment, followed by a three-week interval before repeated medication, with the treatment repeated for a total of at least three cycles plus continuous androgen deprivation therapy. All patients will undergo radical prostatectomy within 3 weeks (±7 days) after the end of treatment.

ELIGIBILITY:
Inclusion Criteria：

① Aged ≥ 18 years and ≤ 85 years;

* Histologically or cytologically confirmed prostate cancer;

  * Patients meeting any of the following disease staging criteria:

    1. Localized high-risk/very high-risk prostate cancer: meeting at least one of the following characteristics (clinical stage T3-T4, Gleason score ≥ 8, primary Gleason pattern 5, or PSA > 20 ng/mL), with no local lymph node metastasis (N0) and no distant metastasis (M0);
    2. Prostate cancer with local lymph node metastasis: presence of local lymph node metastasis (N1) but no distant metastasis (M0);
    3. Metastatic prostate cancer: confirmed as metastatic prostate cancer by imaging examinations; ④ Physical status: Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1; ⑤ Informed consent: All patients voluntarily sign the informed consent form and can adhere to treatment and follow-up.

       Exclusion Criteria：

       ① Any previous or ongoing prostate cancer treatment, including radiotherapy, chemotherapy, androgen deprivation therapy (ADT), etc.;
* A history of previous prostatectomy;

  * Any other severe underlying medical, psychiatric, or psychological diseases that, in the investigator's judgment, may affect the treatment;

    * A history of allergy to the drugs used in the study; ⑤ Refusal to undergo radical prostatectomy; ⑥ Ineligibility to participate in this clinical trial as judged by the investigator.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
pCR or MRD rate | Within three weeks after the operation
PSA response rate | Within one week after the completion of the last treatment cycle (each treatment cycle lasts approximately 25 days)
Biochemical Progression-Free Survival (bPFS) after radical prostatectomy | From the date of random grouping to the date when progression was first recorded or the date of any cause of death (whichever comes first), an assessment was conducted for a period of up to 5 years.

SECONDARY OUTCOMES:
Pathological response after radical prostatectomy (including positive surgical margins, tumor size, extraprostatic extension, seminal vesicle invasion, and lymph node involvement) | Within one month after the surgery
Changes in radiological TNM staging from post-neoadjuvant therapy to pre-surgery | Within one month after the surgery
Other progression-free survival (progression includes radiological progression, castration resistance, need for further therapeutic intervention, etc.) | From the date of random grouping to the date when progression was first recorded or the date of any cause of death (whichever comes first), an assessment was conducted for a period of up to 5 years.
Safety indicator: CTCAE 5.0 Adverse Event Grading | From the date of random grouping to the date when progression was first recorded or the date of any cause of death, an assessment was conducted for a period of up to 5 years.
Quality of life score: EORTC QLQ-C30 scale | From the date of random grouping to the date when progression was first recorded or the date of any cause of death, an assessment was conducted for a period of up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Physician, Study Director — Vice President of Zhongda Hospital Affiliated to Southeast University
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No